CLINICAL TRIAL: NCT01679600
Title: Cardiovascular Rehabilitation Early After Stroke Using Feedback-controlled Robotics-assisted Treadmill Exercise: A Randomised Controlled Pilot Trial
Brief Title: Cardiovascular Rehabilitation Early After Stroke Using Feedback-controlled Robotics-assisted Treadmill Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bern University of Applied Sciences (Other)
Collaborators: Maastricht University (Other); Reha Rheinfelden (Other); Swiss Federal Institute of Technology (Other)
Responsible Party: Principal Investigator, Oliver Stoller, cand. PhD, Bern University of Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CardioRobot
Record Dates: First submitted 2012-08-29; First posted 2012-09-06 (Estimated); Results first posted 2015-08-05 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-07

CONDITIONS: Stroke; Cardiovascular Diseases
Keywords: Rehabilitation; Robotics-assisted Treadmill Exercise; Aerobic Capacity; Exercise Testing
MeSH Terms: conditions — Stroke; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FC-RATE (Experimental): Feedback-controlled robotics-assisted treadmill exercise
  Interventions: Device: Feedback-controlled robotics-assisted treadmill exercise
- RATE (Active Comparator): Robotics-assisted treadmill exercise
  Interventions: Device: Robotics-assisted treadmill exercise

INTERVENTIONS:
Device: Feedback-controlled robotics-assisted treadmill exercise — Progressive cardiovascular exercise using feedback-controlled robotics-assisted treadmill exercise. The first training session is defined to start at 40% of peak work rate (determined from a previous exercise test) to approach 40% of heart rate reserve (Borg scale approximately 11-14). The intensity will then be adjusted on the basis of continuous heart rate data and rating of perceived exertion indications by modulating the target work rate in 5% increments for every subsequent session to reach the target intensity. The target heart rate is set at 40% to 70% of heart rate reserve.
  Other Names: Lokomat system (Hocoma AG, Volketswil, Switzerland)
  Arms: FC-RATE
Device: Robotics-assisted treadmill exercise — Conventional robotics-assisted treadmill exercise, where therapists focus on gait quality only.
  Other Names: Lokomat system (Hocoma AG, Volketswil, Switzerland)
  Arms: RATE

SUMMARY:
The propose of this study is to evaluate the feasibility and the clinical efficiency of feedback-controlled robotics-assisted treadmill exercise (RATE) technology for cardiovascular rehabilitation early after stroke. The investigators hypothesize that feedback-controlled RATE might be suitable and effective to improve cardiovascular fitness and functional carryover in non-ambulatory individuals with sub-acute stroke.

DETAILED DESCRIPTION:
For detailed info: Stoller O, de Bruin ED, Schuster-Amft C, Schindelholz M, de Bie RA, Hunt KJ. Cardiovascular rehabilitation soon after stroke using feedback-controlled robotics-assisted treadmill exercise: study protocol of a randomized controlled pilot trial. Trials. 2013 Sep 22;14(1):304.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of an initial supratentorial stroke
* ≤20 weeks post stroke at intervention onset
* Age ≥18 years
* Functional Ambulation Category (FAC) ≤3
* Ability to understand the procedures and provide informed consent

Exclusion Criteria:

* Contraindications for exercise testing outlined by American College of Sports Medicine (ACSM)
* Contraindications for RATE according to the manufacturer
* Concurrent neurological disease
* Concurrent pulmonary disease
* History of dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rob A. de Bie, Prof., Study Director — Department of Epidemiology, Maastricht University and Caphri Research School, Maastricht, Netherlands; Kenneth J. Hunt, Prof., Study Director — Institute for Rehabilitation and Performance Technology, Bern University of Applied Sciences, Burgdorf, Switzerland; Eling D. de Bruin, PD Dr., Study Director — Institute of Human Movement Sciences and Sport, ETH Zurich, Switzerland; Thierry Ettlin, Prof., Principal Investigator — Reha Rheinfelden, Rheinfelden, Switzerland
Locations (1):
- Reha Rheinfelden, Rheinfelden, Canton of Aargau, Switzerland

REFERENCES:
- [Background] Stoller O, de Bruin ED, Knols RH, Hunt KJ. Effects of cardiovascular exercise early after stroke: systematic review and meta-analysis. BMC Neurol. 2012 Jun 22;12:45. doi: 10.1186/1471-2377-12-45. PMID 22727172
- [Background] Stoller O, Schindelholz M, Bichsel L, Schuster C, de Bie RA, de Bruin ED, Hunt KJ. Feedback-controlled robotics-assisted treadmill exercise to assess and influence aerobic capacity early after stroke: a proof-of-concept study. Disabil Rehabil Assist Technol. 2014 Jul;9(4):271-8. doi: 10.3109/17483107.2013.785038. Epub 2013 Apr 18. PMID 23597319
- [Background] Stoller O, de Bruin ED, Schindelholz M, Schuster C, de Bie RA, Hunt KJ. Evaluation of exercise capacity after severe stroke using robotics-assisted treadmill exercise: a proof-of-concept study. Technol Health Care. 2013;21(2):157-66. doi: 10.3233/THC-130730. PMID 23510976
- [Background] Stoller O, de Bruin ED, Schuster-Amft C, Schindelholz M, de Bie RA, Hunt KJ. Cardiovascular rehabilitation soon after stroke using feedback-controlled robotics-assisted treadmill exercise: study protocol of a randomised controlled pilot trial. Trials. 2013 Sep 22;14:304. doi: 10.1186/1745-6215-14-304. PMID 24053609
- [Result] Stoller O, de Bruin ED, Schindelholz M, Schuster-Amft C, de Bie RA, Hunt KJ. Efficacy of Feedback-Controlled Robotics-Assisted Treadmill Exercise to Improve Cardiovascular Fitness Early After Stroke: A Randomized Controlled Pilot Trial. J Neurol Phys Ther. 2015 Jul;39(3):156-65. doi: 10.1097/NPT.0000000000000095. PMID 26050073
- See also: Institute for Rehabilitation and Performance Technology — http://irpt.ti.bfh.ch
- See also: Reha Rheinfelden — http://www.reha-rheinfelden.ch/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 6 subjects dropped out before assiggnment (abnormal gait pattern due to uncontrollable spasticity, tibia skin lesion due to inadequate padding during familiarization, lack of motivation to produce maximal work rate values, severe groin pain caused by the body weight support harness, suspected cerebrospinal fluid leak, acute respiratory infection)
Groups:
- FC-RATE: Feedback-controlled robotics-assisted treadmill exercise
  Feedback-controlled robotics-assisted treadmill exercise: Human-in-the-loop feedback system to control individual's active work rate
- RATE: Robotics-assisted treadmill exercise
  Robotics-assisted treadmill exercise: Conventional robotics-assisted treadmill exercise
Period: Overall Study
Arm/Group | FC-RATE | RATE
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FC-RATE | RATE | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (12) | 63 (13) | 61 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 3 | 6 | 9
Region of Enrollment [Number; unit: participants]
  Switzerland | 7 | 7 | 14
Type of stroke: ischemic/hemorrhagic [Number; unit: participants]
  ischemic | 5 | 7 | 12
  hemorrhagic | 2 | 0 | 2
Hemiparetic side: right/left [Number; unit: participants]
  right | 5 | 2 | 7
  left | 2 | 5 | 7
Functional Ambulation Classification (0-5) [Mean (Standard Deviation); unit: units on a scale] — Patients will be rated on the following 6 categories: 0: Patient cannot walk, or needs help from 2 or more persons. 1: Patients needs firm continuous support from 1 person who helps carrying weight and with balance. 2: Patient needs continuous or intermittent support of one person to help with balance and coordination. 3: Patient requires verbal supervision or stand-by help from one person without physical contact. 4: Patient can walk independently on level ground, but requires help on stairs, slopes or uneven surfaces. 5: Patient can walk independently anywhere.
  units on a scale | 1 (0.8) | 0.9 (1) | 1 (0.8)
Time poststroke [Mean (Standard Deviation); unit: days] | 52 (42) | 45 (30) | 52 (31)

OUTCOME MEASURES:

1. Primary Outcome: Peak Oxygen Uptake (V'O2peak)
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | FC-RATE | RATE
Number analyzed (Participants) | 7 | 7
mL/min | 1461 (683) | 1494 (672)
Statistical Analysis 1: Comparison: FC-RATE vs RATE; Test type: Superiority or Other; p = 0.53, F1-LD-F1 model by Brunner and Langer

ADVERSE EVENTS:
Time Frame: 10/01/2012-03/31/2014
Arm/Group | FC-RATE | RATE
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes